CLINICAL TRIAL: NCT04580381
Title: Real World Effectiveness of Natalizumab Extended Interval Dosing in Relapsing-Remitting Multiple Sclerosis in a French Cohort
Brief Title: Real World Effectiveness of Natalizumab Extended Interval Dosing in a French Cohort
Acronym: RELEVANT
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: FRA-TYS-19-11504
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2020-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Natalizumab; Extended Interval Dosing
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standard Interval Dosing (SID): Patients continuing Natalizumab treatment with standard interval dosing defined as > 11 infusions per year
  Interventions: Drug: Natalizumab Injection [Tysabri]
- Extended Interval Dosing (EID): Patients switching to extended interval dosing defined as ≤ 10 infusions per year
  Interventions: Drug: Natalizumab Injection [Tysabri]

INTERVENTIONS:
Drug: Natalizumab Injection [Tysabri] — Natalizumab infusion interval according to local practice defining the patient's group

SUMMARY:
Natalizumab (NTZ) use in Multiple Sclerosis (MS) in highly active patients has been largely established during the last Rationale 10 years in both clinical trials and real-world practice. Along with its efficacy, NTZ use has been limited by potential risk of progressive multifocal leukoencephalopathy (PML). Thus, several studies have tried to assess how to minimize this risk.

One suggested approach is to move from the standard interval dose (SID) of 4 weeks to an extended interval dose (EID) of 5 weeks or longer. Extending the dosing interval of NTZ has been practiced by some physicians with the intention of improving the benefit/risk of the treatment by reducing the exposure-dependent risk of progressive multifocal leukoencephalopathy (PML) while maintaining efficacy. We propose to retrospectively analyze data from clinical records coming from RRMS patients treated in France at 5 different centers; Caen, Nice, Bobigny and Toulouse hospitals as well as Percy Military Hospital, to evaluate the effectiveness of natalizumab EID in subjects who have previously been treated with natalizumab SID for 12 months, in relation to continued SID treatment. In the clinical practice of these centers, patients are shifted after minimum 12 months under SID to an EID of 6 weeks regardless antibody JC serum status. Clinical, magnetic resonance imaging (MRI) and serum anti-JCV antibody status data are collected when available.

The objective of this study is to assess the efficacy in term of ARR and safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving at least 11 infusions of natalizumab as disease-modifying monotherapy for RRMS that is consistent with the approved dosing

Exclusion Criteria:

* Patients for whom the NTZ infusion history and/or MRI and clinical history is not available.
* Patients with dosing gap defined as >=12 weeks between any two doses.
* Patients with over dose defined as <3 weeks between any two doses.
* Pregnancy during the follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving Natalizumab as disease-modifying monotherapy for RRMS
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Annualized Relapse Ratio | baseline to 12 month follow-up
  relapse rate per patient per year

SECONDARY OUTCOMES:
Disability progression | baseline to 12 month follow-up
  Increase in EDSS score during the follow-up period
NEDA-3 achievement | baseline to 12 month follow-up
  Estimation of the proportion of patients achieving NEDA-3 criteria at the end of the follow-up period
Radiological activity | baseline to 12 month follow-up
  Detection of increase MRI activity defined as new or enlarged T2 lesions and/or new gadolinium enhancing lesions

OTHER OUTCOMES:
Safety outcome | baseline to 12 month follow-up
  Description of PML cases and variations in anti-JCV antibody status when available

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Department of Neurology, CHU Bobigny-Avicenne, Bobigny
  - Department of Neurology, CHU de Caen, Caen
  - Department of Neurology, Percy Military Hospital, Clamart
  - Department of Neurology, CHU Nice, Nice
  - Department of Neurology, CHU Toulouse Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pelle J, Briant AR, Branger P, Derache N, Arnaud C, Lebrun-Frenay C, Cohen M, Mondot L, De Seze J, Bigaut K, Collongues N, Kremer L, Ricard D, Bompaire F, Ohlmann C, Sallansonnet-Froment M, Ciron J, Biotti D, Pignolet B, Parienti JJ, Defer G. Real-World Effectiveness of Natalizumab Extended Interval Dosing in a French Cohort. Neurol Ther. 2023 Apr;12(2):529-542. doi: 10.1007/s40120-023-00440-5. Epub 2023 Feb 10. PMID 36763307